CLINICAL TRIAL: NCT04188444
Title: Thrombotic Profile of Ovarian Stimulation Protocols in Reproductive Medical Assistance: a Prospective Cohort Study
Brief Title: Prothrombotic Biomarkers and Ovarian Stimulation
Acronym: HEMOSTIM
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Casini Alessandro, Principal Investigator, University Hospital, Geneva
Other Study IDs: CCER2019-02134
Record Dates: First submitted 2019-11-27; First posted 2019-12-05 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Sterility, Female; Reproductive Technology, Assisted
Keywords: Ovarian stimulation; thrombin generation; haemostasis; thrombosis
MeSH Terms: conditions — Infertility, Female; Helping Behavior; Thrombosis | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Agonist: Ovarian stimulation with agonist of GnRH
  Interventions: Biological: Blood test
- Antagonist: Ovarian stimulation with antagonist of GnRH
  Interventions: Biological: Blood test

INTERVENTIONS:
Biological: Blood test — 20 ml of blood, three times

SUMMARY:
The aim of this study is to assess the impact of different protocols used for ovarian stimulation during in vitro fertilization procedures (IVF) on prothrombotic biomarkers (blood coagulation markers associated with thromboembolic events) in the units of reproductive medicine in two university hospitals (HUG, Geneva and CHUV, Lausanne).

DETAILED DESCRIPTION:
HEMO-STIM is a prospective multicentric cohort study of subfertile women undergoing ART. It is an epidemiologic observational study. All women older than 18 years attending the reproductive medicine unit (UMREG, Geneva, HUG or UMR, Lausanne, CHUV) and undergoing an IVF have been and will be recruited consecutively and included. The type of stimulation protocol used is recorded.

All measurements (specific haemostasis test with a thrombin generation assay before and after adjunction of APC) that are part of the study will be performed in the HUG laboratories in order to limit inter-dosage variability.

The 1st blood test will be performed at inclusion in the absence of any hormonal treatment (T1). A 2nd blood test will be performed on the day of ovulation triggering (T2). A 3rd blood test will be performed 7 days after ovulation triggering (T3).

The comparison of different protocols has never been performed and data on the effect of antagonist protocols for IVF on haemostasis are lacking. The measurement of intermediate biomarkers of thromboembolic risk during different IVF stimulation protocols (agonists and antagonists) would allow the comparison of their thrombotic profile and to optimize the risk/benefit ratio during ART by prescribing protocols at lower vascular risk, in particular in women identified as being at risk for thromboembolic events.

ELIGIBILITY:
Inclusion Criteria:

* Women older than 18 years
* Sub-fertile and undergoing IVF

Exclusion Criteria:

* >43 years old

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women will be recruited in reproductive unit from 2 hospitals (HUG, Geneva and CHUV, Lausanne) in Switzerland
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Change in normalized APC sensitivity ratio | T1: inclusion; T2: day1 ovarian stimulation; T3: day7 after ovarian stimulation
  Haemostasis parameters: thrombin Generation Assay

SECONDARY OUTCOMES:
Change in fibrinolysis assay | T1: inclusion; T2: day1 ovarian stimulation; T3: day7 after ovarian stimulation
  haemostasis parameters: turbidimetry assay

CONTACTS AND LOCATIONS:
Overall Officials: Justine Hugon-Rodin, MD, PHD, Principal Investigator — Hôpitaux de Paris, Université de Paris; Alessandro Casini, MD, Principal Investigator — University Hospital, Geneva
Locations (2):
- Switzerland (2):
  - University Hospitals of Geneva, Geneva
  - CHUV, Lausanne

REFERENCES:
- [Derived] Hugon-Rodin J, Casini A, Benard J, Poncet A, Raverot V, Fontana P, Vulliemoz N, Streuli I. Prothrombotic biomarkers during controlled ovarian stimulation for assisted reproductive technology. Fertil Steril. 2023 Jun;119(6):976-984. doi: 10.1016/j.fertnstert.2023.02.009. Epub 2023 Feb 16. PMID 36805437